CLINICAL TRIAL: NCT07180940
Title: Comparison of Perineural Dexamethasone Versus Dexmedetomidine as Adjuvants to Erector Spinae Plane Block in Lumbar Spine Surgery: A Randomized, Double-blind, Controlled Trial
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01/2025
Record Dates: First submitted 2025-09-12; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Spine Disease; Spinal Diseases
MeSH Terms: conditions — Spinal Diseases | interventions — Sodium Chloride; Dexamethasone; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Placebo Comparator): Bilateral ESPB (2 x 20ml 0.2% ropivacaine with 1ml 0.9% NaCl)
  Interventions: Drug: 0.9%NaCl
- Dexamethasone group (Experimental): Bilateral ESPB (2 x 20ml 0.2% ropivacaine with 2mg dexamethasone)
  Interventions: Drug: Dexamethasone 4mg
- Dexmedetomidine group (Experimental): Bilateral ESPB (2 x 20ml 0.2% ropivacaine with 25ug dexmedetomidine)
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: 0.9%NaCl — 2 x 20ml 0.2% ropivacaine with 2ml of 0.9% NaCl
  Arms: Control group
Drug: Dexamethasone 4mg — 2 x 20ml 0.2% ropivacaine with 2mg of dexamethasone
  Arms: Dexamethasone group
Drug: Dexmedetomidine — 2 x 20ml 0.2% ropivacaine with 25ug Dexmedetomidine
  Arms: Dexmedetomidine group

SUMMARY:
This clinical study aims to determine which of two medications-dexamethasone or dexmedetomidine-works better and is safer when used together with a local anesthetic (ropivacaine) in a type of nerve block called the erector spinae plane block (ESPB). This block helps reduce pain after lumbar spine surgery.

DETAILED DESCRIPTION:
All participants will receive general anesthesia for surgery and, in addition, a nerve block on both sides of the lower back. The nerve block will be done with ultrasound guidance and will include ropivacaine plus either dexamethasone or dexmedetomidine. Patients will be randomly assigned to one of these two groups, and neither the patient nor the doctors checking pain after surgery will know which medication was used.

The main goal is to see how much opioid pain medicine patients need during the first 24 and 48 hours after surgery. Other things we will look at include how strong the pain is, how soon pain relief is necessary, if there are any side effects like nausea or low blood pressure, and if there are any complications related to the block.

This study will help doctors choose the best option to manage pain after spine surgery while reducing the need for opioids and their side effects.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to N/A (no limit)
* Scheduled for elective lumbar spine surgery (e.g., decompression or fusion) via posterior approach
* American Society of Anesthesiologists (ASA) physical status I-III
* Body weight ≥ 50 kg
* Ability to provide written informed consent
* Expected postoperative hospitalization of at least 48 hours

Exclusion Criteria:

* Known allergy or contraindication to ropivacaine, dexamethasone, or dexmedetomidine
* Infection at or near the site of block placement
* Coagulation disorders or current use of anticoagulant therapy (not discontinued per guidelines)
* Chronic opioid use or opioid dependence
* Neurological or psychiatric disorders interfering with pain assessment
* Diabetes mellitus with poorly controlled glycemia (e.g., HbA1c > 8%)
* Severe hepatic or renal dysfunction
* Body mass index (BMI) > 40 kg/m²
* Pregnancy or breastfeeding
* Refusal or inability to cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total opioid Consuption | 48 hours after surgery
  Cumulative opioid consumption during the first 24 and 48 hours after surgery, converted to morphine milligram equivalents (MME)

SECONDARY OUTCOMES:
NRS | 4 hours after surgery
  Numerical Rating Scale (0 - no pain; 10 - the worst pain ever)
NRS | 8 hours after surgery
  Numerical Rating Scale (0 - no pain; 10 - the worst pain ever)
NRS | 12 hours after surgery
  Numerical Rating Scale (0 - no pain; 10 - the worst pain ever)
NRS | 24 hours after surgery
  Numerical Rating Scale (0 - no pain; 10 - the worst pain ever)
NRS | 48 hours after surgery
  Numerical Rating Scale (0 - no pain; 10 - the worst pain ever)
Nerve injury | 12 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve injury | 24 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
Nerve injury | 48 hours after surgery
  Nerve damage assesment will be performed using the nerve damage score (N0- no nerve damage; N1- minor - sensory paresthesia; N2- major -complete sensory anesthesia; N3- Complete- complete motor defect with or without paraesthesia; N4-CRPS- Complex Regional Pain Syndrome)
adverce effects | 48 hours after surgery
  nausea, vomitting, bradycardia, hypotension
Time to first rescue analgesia | 48 hours after surgery
  Time after surgery when the patient needs rescue analgesia for the first time
blood glucose | 12 hours after surgery
  Blood glucose concentration measured postoperatively
blood glucose | 24 hours after surgery
  Blood glucose concentration measured postoperatively
blood glucose | 48 hours after surgery
  Blood glucose concentration measured postoperatively
NLR - Neutrophil-to-Lymphocyte Ratio | 12 hours after surgery
  NLR will be calculated from complete blood count results
NLR - Neutrophil-to-Lymphocyte Ratio | 24 hours after surgery
  NLR will be calculated from complete blood count results
NLR - Neutrophil-to-Lymphocyte Ratio | 48 hours after surgery
  NLR will be calculated from complete blood count results
PLR - Platelet-to-Lymphocyte Ratio | 12 hours after surgery
  PLR will be calculated from complete blood count results
PLR - Platelet-to-Lymphocyte Ratio | 24 hours after surgery
  PLR will be calculated from complete blood count results
PLR - Platelet-to-Lymphocyte Ratio | 48 hours after surgery
  PLR will be calculated from complete blood count results

CONTACTS AND LOCATIONS:
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poland

IPD SHARING:
Plan to Share IPD: Yes